CLINICAL TRIAL: NCT05588960
Title: Investigating Cerebral Oxygenation in the Newborn: An Observational Study Investigating Cerebral Oxygenation in Newborn Infants at High Risk of Brain Injury
Brief Title: Investigating Cerebral Oxygenation in the Newborn
Acronym: ICON
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Prism Training and Consultancy (Unknown); Simpsons Special Care Babies (Unknown)
Responsible Party: Sponsor
Other Study IDs: AC22120
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn; Neonatal Encephalopathy; Premature Infant Disease
Keywords: Spectroscopy, near infrared; Cerebral oxygenation; Cerebral haemodynamics; Newborn brain injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Term/Near-Term Group: Cohort of term/near-term infants undergoing therapeutic hypothermia for moderate to severe HIE. Data collected from NIRS monitoring and other assessments/investigations that are part of routine clinical care. There are no additional study specific interventions or exposures for this group.
- Preterm Group (Sub-study 1, First 72 hours after birth): Cohort of infants born at less than 28 weeks gestational age. Data collected from NIRS monitoring, other physiological monitoring, cranial ultrasound scans and neurodevelopmental follow up assessments that are part of routine clinical care. This data will be analysed to fulfil secondary study objectives. There are no additional study specific interventions or exposures for this group.
- Preterm Group (Sub-study 2, Skin-to-skin care): Cohort of infants born at less than 28 weeks gestational age who are considered by clinical team to be suitable to undergo period of skin-to-skin care. Participants will undergo additional research-specific period(s) of NIRS monitoring before, during and after period(s) of skin-to-skin care. Participants with and without severe brain injury on cranial ultrasound will be recruited to allow comparison.
  Interventions: Device: Near-infrared spectroscopy monitoring (Masimo O3 Regional Oximeter with Neonatal Sensor)
- Preterm Group (Sub-study 3, Bronchopulmonary dysplasia): Cohort of infants born at less than 28 weeks gestational age who will undergo an additional research-specific period of NIRS monitoring at 36 weeks corrected gestational age. Participants with and without bronchopulmonary dysplasia (BPD) will be recruited to allow comparison.
  Interventions: Device: Near-infrared spectroscopy monitoring (Masimo O3 Regional Oximeter with Neonatal Sensor)

INTERVENTIONS:
Device: Near-infrared spectroscopy monitoring (Masimo O3 Regional Oximeter with Neonatal Sensor) — Masimo O3 neonatal sensor will be applied:
  * At least 30 minutes before a period of skin-to-skin care with a caregiver commences (baseline condition).
  * Throughout the period of skin-to-skin care, which should continue for a minimum of 1 hour.
  * For at least 1 hour after the participant is returned to their incubator (post-intervention condition).
  The protocol accounts for a 30 minute washout period between each study epoch. Therefore, at least 30 minutes of study data will be collected for each epoch.
  Groups: Preterm Group (Sub-study 2, Skin-to-skin care)
Device: Near-infrared spectroscopy monitoring (Masimo O3 Regional Oximeter with Neonatal Sensor) — Masimo O3 neonatal sensor will be applied:
  ▪ For 24 hours once the participant reaches 36 weeks corrected gestational age.
  Groups: Preterm Group (Sub-study 3, Bronchopulmonary dysplasia)

SUMMARY:
The goal of this single centre observational study is to use near-infrared spectroscopy (NIRS) monitoring to investigate cerebral oxygenation in two groups of newborn infants who are at high risk of brain injury. The NIRS monitor used in this study will be the Masimo O3 regional oximeter with neonatal sensors.

Near-infrared spectroscopy (NIRS) monitoring uses near-infrared light to measure oxygen levels in the brain tissue (cerebral oxygenation). It provides information about blood flow to the brain and the balance between oxygen supply and demand in the brain tissue. It is non-invasive, safe and used routinely to monitor term and premature babies in the neonatal intensive care unit (NICU).

This study will recruit two groups of infants admitted to the NICU who are at risk of brain injury in the newborn period, namely:

* Term and near-term babies who are undergoing cooling treatment (therapeutic hypothermia) for moderate to severe hypoxic ischaemic encephalopathy (HIE).
* Preterm babies who are born extremely prematurely (before 28 weeks of pregnancy).

In the term/near-term group, the primary aims of the study are:

* To investigate if cerebral oxygenation during and after cooling treatment relates to markers of brain injury detected on detailed brain scans (MRI and MRS scans).
* To describe any changes in cerebral oxygenation which occur during and after seizures (fits) in babies undergoing cooling treatment.

In the preterm group, the primary aims of the study are:

* To investigate if any changes in cerebral oxygenation occurring during skin-to-skin care are different in premature babies with brain injury (bleeding or cysts in the brain seen on ultrasound scan) compared to babies without these changes.
* To investigate if cerebral oxygenation at 36 weeks corrected gestational age differs in babies with bronchopulmonary dysplasia (BDP, a chronic lung disease of prematurity) compared to babies without BPD.

DETAILED DESCRIPTION:
TERM/NEAR-TERM GROUP

Hypoxic-ischaemic encephalopathy (HIE) is the most common cause of newborn brain injury in term and near-term infants. It is caused by a lack of oxygen supply or blood flow to the brain around the time of delivery. It is classified as mild, moderate or severe based on the symptoms present. Babies with moderate or severe HIE are treated with 3 days of cooling treatment (therapeutic hypothermia). This treatment protects the brain and reduces the risk of death or disability. However, despite this treatment some babies do not survive or develop life-long disabilities. Therefore, research into potential new treatments for HIE is ongoing.

Currently, the best tests available to detect brain injury and predict later outcome are magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) scans of the brain. However, these are only performed after therapeutic hypothermia is complete, between 5 to 15 days after birth. It would be advantageous if there was a tool that could identify brain injury earlier in the course, as this could facilitate identification of babies who may benefit most from new treatments in the future. Brain injury due to HIE can cause altered blood flow and oxygen levels in the brain, which can be detected by NIRS monitoring. Therefore, it is possible that NIRS monitoring could facilitate earlier detection of brain injury in this group. To understand this further, it is essential to further investigate the relationship between cerebral oxygenation measurements derived by NIRS monitoring and current markers of brain injury. Therefore, the first research question in this group is:

▪ How does cerebral oxygenation during and after therapeutic hypothermia (TH) for moderate to severe HIE relate to markers of brain injury detected on MRI and MRS scans performed between 5 to 15 days after birth?

Seizures are common in babies with HIE. Frequent or prolonged seizures are associated with higher risk of adverse outcomes. It is possible that seizures contribute to on-going injury to the brain due to disrupting the balance of oxygen supply and demand in the brain. This study aims to understand more about this by answering the following research question:

▪ How does cerebral oxygenation change during seizures in infants undergoing therapeutic hypothermia for moderate to severe HIE?

In this group, NIRS monitoring is used routinely in the study centre for all infants undergoing therapeutic hypothermia. Therefore, data from routine NIRS monitoring alongside other data collected as part of routine clinical care (clinical assessments, aEEG and MRI/MRS) will be analysed in a novel way to answer the research questions.

Routinely acquired clinical data will also be analysed to meet the following secondary objectives:

* To assess the predictive value of mean cerebral oxygenation at each pre-defined time point as a marker for brain injury detected on MRI/MRS and to suggest optimal cut-offs for predicting brain injury at each time point if applicable.
* To compare any changes in cerebral oxygenation occurring in association with seizures occurring in infants with brain injury detected on MRI/MRS scans to those without brain injury on MRI/MRS scans.
* To compare mean cerebral oxygenation at pre-specified time points during and after therapeutic hypothermia to outcomes of neurodevelopmental assessments in infancy and at the age of 2 years.

PRETERM GROUP

Although survival of infants born extremely prematurely (before 28 weeks of pregnancy) has improved over recent decades, these babies remain at high risk of neurodevelopmental disabilities due to brain injury or dysmaturation. The immature brain is vulnerable to fluctuations in cerebral blood flow and oxygenation, which may be detected by NIRS monitoring. In this group of infants, recognisable patterns of brain injury include intraventricular haemorrhage (bleeding into the fluid filled spaces in the brain) and periventricular leukomalacia (cysts in the brain tissue). These conditions can be detected by ultrasound scans of the brain which are performed routinely for all premature babies.

Skin-to-skin care, when an infant is nursed in direct skin-to-skin contact with a parent or carer, is commonly undertaken in the neonatal intensive care unit. There are many documented benefits for babies and their parents. Previous studies have investigated cerebral oxygenation during skin-to-skin care, however, these studies have not included infants with severe brain injury. This study seeks to understand whether more severe patterns of brain injury detected on cranial ultrasound affects cerebral oxygenation during skin-to-skin care by answering the following research question:

▪ Do changes in cerebral oxygenation during periods of skin-to-skin care versus flanking periods of incubator care differ in preterm infants with severe brain injury compared to infants without severe brain injury?

Bronchopulmonary dysplasia (BPD) is a chronic lung disease that occurs in premature babies. It is diagnosed if a baby still requires extra oxygen or other breathing support at 36 weeks corrected gestational age (4 weeks before their due date). It is associated with brain dysmaturation and a higher chance of neurodevelopmental disabilities. It is possible that lower cerebral oxygenation levels contribute to brain dysmaturation in this group. Therefore, this study aims to answer the following research question:

▪ Does cerebral oxygenation and cerebral hypoxic burden (a measure of low oxygen levels in the brain accounting for severity and duration) differ in extremely preterm infants with bronchopulmonary dysplasia (BPD) compared to infants without BPD at 36 weeks corrected gestational age?

In the study centre, NIRS monitoring is routine for all infants born at less than 28 weeks for the first 72 hours after birth. Therefore, to answer the above research questions, NIRS monitoring will also be applied for additional periods out with routine clinical care for infants recruited to the study. No other changes to routine clinical care will be made for infants recruited to the study.

Data from routine NIRS monitoring for the first 72 hours after birth and from routine scans and neurodevelopmental follow up assessments will also be collected to fulfil the following secondary objectives:

▪ To compare cerebral oxygenation and cerebral hypoxic burden over the first 72 hours after birth to: worst grade of injury detected on routine screening cranial ultrasound scans and outcomes of neurodevelopmental assessments in infancy and at the age of 2 years.

ELIGIBILITY:
TERM/NEAR-TERM GROUP

INCLUSION CRITERIA:

1. Infants born at greater than or equal to 34 weeks gestational age undergoing therapeutic hypothermia as an intervention for moderate to severe neonatal encephalopathy. These infants will meet the following criteria for treatment:

   * Evidence of intrapartum asphyxia as defined by ANY of the following features: Apgar score of 5 or less at 10 minutes after birth; ongoing need for endotracheal or mask ventilation at 10 minutes after birth; pH <7.00 in cord or baby sample within 60 minutes of birth; base deficit greater than or equal to 16mmol/L in cord or baby sample within 60 minutes of birth.
   * Moderate or severe encephalopathy, including ALL of the following criteria OR altered consciousness plus seizures: altered consciousness (reduced or absent response to stimulation); abnormal primitive reflexes (weak or absent suck or Moro response); abnormal tone (hypotonia, flaccid).
2. Signed parental consent form.

EXCLUSION CRITERIA:

1. Lack of signed parental consent form and/or parental decision not to participate.
2. Infants with life threatening congenital malformations.
3. Infants with encephalopathy caused by differing pathology to hypoxia-ischaemia.

PRETERM GROUP

INCLUSION CRITERIA:

1. Infants born at less than 28 weeks completed gestation.
2. Signed informed parental consent form for each specific section/sub-study.
3. For skin-to-skin sub-study: considered by responsible clinical team to be eligible for skin-to-skin care as per usual local practice.
4. For BPD sub-study: infants born at less than 28 weeks gestational age surviving to 36 weeks corrected gestational age. Infants with and without a diagnosis of BPD will be recruited to allow for comparison of cerebral oxygenation between these groups.

EXCLUSION CRITERIA:

1. Lack of signed parental consent form and/or parental decision not to participate.
2. Decision not to provide active (survival focussed) neonatal management.
3. Infants with life threatening congenital malformation.
4. Infants in whom there is a particularly high level of concerns regarding skin fragility or loss of skin integrity resulting in application of NIRS probe being contraindicated.
5. Infants who are transferred back to local centres will be excluded from the BPD sub-study if transferred back to local centre prior to 36 weeks corrected gestational age and from follow-up data collection due to difficulties achieving acquisition of full data set for babies followed up in health boards outwith NHS Lothian.

Ages: 1 Day to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit a cohort of term/near-term and preterm infants who admitted to the neonatal intensive care unit at the Simpson Centre for Reproductive Health (Edinburgh, NHS Lothian, UK) and are at risk of brain injury or brain dysmaturation.
  Potential participants will be identified through admission to the neonatal intensive care unit. Once eligibility is confirmed, a member of the research team will approach parents to discuss the study and invite the baby to enter the study.
  Participants will be recruited over a 2 year period.
  Preterm infants may be enrolled in more than one sub-study should their parents provide informed consent for this.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Term/Near-Term Group: Primary Outcome 1 | Birth-15 days
  Mean cerebral oxygenation calculated over 1 hour periods at pre-defined time points during therapeutic hypothermia and after completion of rewarming compared to presence/absence of brain injury on magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) performed between 5-15 days after birth.
  Brain injury will be defined as:
  * NICHD NRN MRI score of ≥2A
  * Lactate to n-acetylaspartate peak ratio of >0.39 on MRS
Term/Near-Term Group: Primary Outcome 2 | Birth-5 days
  Maximum change in cerebral oxygenation from baseline occurring during electrical seizures detected on aEEG and cerebral hypoxic burden (expressed in % hours) for any periods of cerebral hypoxia associated with seizures.
Preterm Group - Skin-to-skin sub-study: Primary Outcomes | 2.5 hours
  Change in mean cerebral oxygenation (calculated every 5 minutes) and in variability of cerebral oxygenation during a period of skin-to-skin care compared to periods of incubator care before (pre-intervention) and after (post-intervention) skin-to-skin care.
  These measures will be compared in infants with and without severe brain injury detected on routine cranial ultrasound scans. Severe brain injury will be defined as:
  * Grade III or IV intraventricular haemorrhage
  * Cystic periventricular leucomalacia
Preterm Group - BPD sub-study: Primary Outcomes | 24 hours
  Mean cerebral oxygenation measured over a 24-hour period at 36 weeks corrected gestational age and cerebral hypoxic burden (expressed in % hours) of any periods of cerebral hypoxia over this 24-hour epoch.
  These measures will be compared in infants with and without a diagnosis of bronchopulmonary dysplasia. Bronchopulmonary dysplasia will be defined as the need for any additional respiratory support (including supplementary oxygen) at 36 weeks corrected gestational age.

SECONDARY OUTCOMES:
Term/Near-Term Group: Secondary Outcome 1 | Birth-12 to 15 weeks
  Outcome of General Movements Assessment at term and between 12 to 15 weeks post-term age. High-risk patterns will be defined as cramped synchronised pattern (term equivalent age) and absent fidgety movements (12-15 weeks post-term).
Term/Near-Term Group: Secondary Outcome 2 | 2 years
  Outcome at 2 years of age. Adverse outcome will be defined as death or moderate-severe neurodevelopmental disability as follows:
  * Moderate: Cerebral palsy with GMFCS level 2; Bayley III composite motor/congitive/language score of <85; hearing impairment without need for amplification; persistent seizure disorder.
  * Severe: Cerebral palsy with GMFCS level ≥3; Bayley III composite motor/cognitive/language score of <70; hearing impairment requiring hearing aids; blindness.
Preterm Group: Secondary Outcome 1 | Birth-max 14 weeks
  Comparison of mean cerebral oxygenation and cerebral hypoxic burden (expressed in % hours) for the first 72 hours after birth to findings of routine cranial ultrasound scans at:
  * 1 day after birth
  * 2 days after birth
  * 3 days after birth
  * 7 days after birth
  * Term equivalent age
Preterm Group: Secondary Outcome 2 | Birth-12 to 15 weeks
  Comparison of mean cerebral oxygenation and cerebral hypoxic burden (expressed in % hours) for the first 72 hours after birth to outcomes of General Movements Assessment at term equivalent age and between 12 to 15 weeks post-term age. High-risk patterns will be defined as cramped synchronised pattern (term equivalent age) and absent fidgety movements (12-15 weeks post-term).
Preterm Group: Secondary Outcome 3 | 2 years
  Comparison of mean cerebral oxygenation and cerebral hypoxic burden (expressed in % hours) for the first 72 hours after birth to outcome at 2 years corrected gestational age. Adverse outcome will be defined as death or moderate-severe neurodevelopmental disability as follows:
  * Moderate: Cerebral palsy with GMFCS level 2; Bayley III composite motor/congitive/language score of <85; hearing impairment without need for amplification; persistent seizure disorder.
  * Severe: Cerebral palsy with GMFCS level ≥3; Bayley III composite motor/cognitive/language score of <70; hearing impairment requiring hearing aids; blindness.

CONTACTS AND LOCATIONS:
Overall Officials: Helen L Turner, MBChB (Hons), Principal Investigator — University of Edinburgh/NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the study and after primary publications by the study team, all collected anonymous IPD will be shared in line with the FAIR principles (findable, accessible, interoperable and resuable). Parents will have the option to opt out of their child's anonymous data being shared for the purposes of further research at the time of consent.
  Data will be made available through DataShare, a data respository run by The University of Edinburgh. This will be maintained indefinitely by the University of Edinburgh Data Library staff. Associated metadata will be created in Pure (the University's Current Research Information System) which will be linked to the dataset in DataShare.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared after primary publications by the study team, which are likely to take 6-12 months after the end of the project.
Access Criteria: When data is deposited in DataShare, a DOI will be acquired. This DOI will be used in all communications regarding the data, for example, publications and presentations. A data access statement will be included in all publications. Data on DataShare will be licensed under a CC BY license.
  A metadata will be created in Pure (the University's Current Research Information System) which will be linked to the dataset in DataShare. Pure metadata records are published to Edinburgh Research Explorer, which provides a searchable public view of the University's research activities.